CLINICAL TRIAL: NCT03965429
Title: Immunological Follow-up After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: SIA-CSH
Status: Active, not recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: INSERM-U1068 (Unknown)
Responsible Party: Sponsor
Other Study IDs: SIA-CSH-IPC 2015-017; 2019-000814-13 (EudraCT Number)
Record Dates: First submitted 2019-05-16; First posted 2019-05-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Malignant Hemopathy
Keywords: malignant hemopathy; allogeneic hematopoietic stem cell transplant; blood collection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Systematic longitudinal collection of blood samples for any patient receiving an allogeneic CSH transplant in our facility, regardless of donor category selected and type of graft used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Donor: In the case of a transplant from an intrafamily donor (genoid or haploid), we will also collect blood samples from the donor.
  Interventions: Other: Blood samples (additional tubes from care) at inclusion
- Receiver: Systematic longitudinal collection of blood samples for any patient receiving an allogeneic CSH transplant in our facility, regardless of donor category selected and type of graft used
  Interventions: Other: Blood samples (additional tubes from care) longitudinal

INTERVENTIONS:
Other: Blood samples (additional tubes from care) longitudinal — Some sampling times will be systematic, while others will only be performed in the presence of specific post-transplant clinical events (eg relapse, GVH ...).
  Groups: Receiver
Other: Blood samples (additional tubes from care) at inclusion — In the case of a transplant from an intrafamily donor (genoid or haploid), we will also collect blood samples from the donor. A single blood sample of 28 mL (7 EDTA tubes) will be made.
  In order not to represent an additional sample for the donor, this sample will be taken before the mobilization of the hematopoietic stem cells, during the biological assessment required for the biological donation qualification.
  Groups: Donor

SUMMARY:
Description of the evolution of the biological characteristics of immune blood populations and biomarkers of interest in patients who have received allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
a more in-depth analysis of the different immune cell sub-populations as well as serum markers (cytokines) would provide a better understanding of post-allograft immune reconstitution mechanisms and identify potential immunologic biomarkers predictive of GVH or relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Allogeneic hematopoietic stem cell transplant for hematological malignancy
2. Patients 18 years of age or older
3. Signed consent to participation
4. Membership in a social security scheme, or beneficiary of such a scheme.

Exclusion Criteria:

* A person of legal age subject to a legal protection measure (major under guardianship, curatorship or court bail), or unable to express consent (language criteria included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is male and / or female over 18 years of age with hematologic malignancies receiving allogeneic hematopoietic stem cell transplantation and corresponding donors.
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the immune blood populations in patients who have received allogeneic hematopoietic stem cell transplantation. | 5 years after HSC transplantation
  longitudinal study of the immune subpopulations of allografted patients for hematological malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Raynier Devillier, MD, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France

IPD SHARING:
Plan to Share IPD: No